CLINICAL TRIAL: NCT02793778
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Effectiveness of a Nutritional Intervention in Improving the Intestinal Mucosal Health Status in Subjects With Crohn's Disease (CD) Receiving Anti-TNF Therapy
Brief Title: Efficacy of CROWN in Repair and Maintenance of the Intestinal Mucosa in Patients With CD Receiving Anti-TNF Therapy
Acronym: PIONEER-CD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: enrollment
Sponsor: Prometheus Laboratories (Industry)
Collaborators: Nestlé Health Science Spain (Industry); Nestec Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13.06.CLI
Record Dates: First submitted 2016-06-01; First posted 2016-06-08 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; mucosal healing; inflammatory bowel disease; Medical Food; Nutritional intervention
MeSH Terms: conditions — Crohn Disease; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Inflammatory Bowel Diseases | interventions — Crowns

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CROWN (Experimental): CROWN: A nutritionally based therapy with a high protein content, formulated as a powder. Twice a day, preferable 1 hour before or more than 2 hours after meals, for up to 24 weeks
  Interventions: Drug: CROWN
- CROWN Placebo (Placebo Comparator): Placebo: An appearance and volume matched formulated powder. Twice a day, preferable 1 hour before or more than 2 hours after meals, for up to 24 weeks
  Interventions: Drug: CROWN Placebo

INTERVENTIONS:
Drug: CROWN — A nutritionally based therapy, formulated as a powder, administered twice a day, preferable 1 hour before or more than 2 hours after meals, for up to 24 weeks
  Arms: CROWN
Drug: CROWN Placebo — Placebo, formulated as a powder, administered twice a day, preferable 1 hour before or more than 2 hours after meals, for up to 24 weeks
  Arms: CROWN Placebo

SUMMARY:
The purpose of this study is to evaluate CROWN's efficacy in supporting the repair and maintenance of the intestinal mucosa of patients with moderately to severely active Crohn's Disease receiving anti-Tumor Necrosis Factor (TNF) therapy (infliximab, adalimumab, certolizumab)

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of an orally administered nutritional intervention (CROWN) in subjects with Crohn's Disease (CD) to support Standard Of Care (SOC) treatment in the repair and maintenance of the intestinal mucosa over a 24 week period. SOC is defined as having been on a stable maintenance dose of an anti-Tumor Necrosis Factor (TNF) agent within 24 weeks of its initiation.

ELIGIBILITY:
Inclusion Criteria:

Crohn's Disease patient who has derived clinical benefit from the Standard of Care therapy, but continues to have evidence of incomplete healing of the intestinal mucosa.

1. Adults (18-85 years of age) with a known history of symptomatic CD confirmed by endoscopy or radiology
2. CDAI score ≤ 350
3. Active endoscopic disease (SES-CD score ≥ 6) documented during the study screening phase or SES-CD score ≥ 4 if isolated ileal disease
4. On a stable dose of infliximab, adalimumab, or certolizumab therapy for 8 weeks prior to randomization as part of SOC
5. Able to consume oral nutrition for up to 24 weeks consisting of two 4 oz (120 ml) servings daily
6. Able to understand the informed consent process, willing to follow study instructions and likely to complete all required visits and procedures, including the use of an electronic device to collect study data, home computer or tablet and internet access to complete online food frequency questionnaire, and undergo 2 endoscopies in a 6 month period

Exclusion Criteria:

Subjects with one or more of the following criteria are excluded from participation in the study:

1. If female, subject is pregnant, nursing, or planning to become pregnant during the study period or is of childbearing potential and unable or unwilling to use a reliable form of contraception during the study
2. Fistula known to be contributing to diarrhea
3. Recent or current history of bowel obstruction
4. Stricturing disease with evidence of bowel dilation proximal to stricture on imaging
5. Anticipated need for gastrointestinal surgical therapy in the next 6 months
6. Current treatment with a systemic corticosteroid at dose greater than 20 mg of prednisone (or equivalent) at screening
7. Change in any antimetabolite therapy within 8 weeks prior to randomization
8. Current treatment with antibiotics for CD (ciprofloxacin, metronidazole) at screening
9. Current ostomy
10. Serious infection, neoplasia or other medical conditions which would interfere with participation in the study, in the opinion of the Investigator
11. Evidence of Clostridium difficile infection in the previous 4 weeks
12. History of non-compliance with clinical protocols
13. Active participation in another CD trial or received an investigational product within the past 4 weeks
14. Diagnosis of celiac disease
15. Known sensitivity to milk or soy protein
16. In the Investigator's opinion, subject has any condition or situation which makes the subject unsuitable for study participation, may put the subject at significant risk, or may confound the study results

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-07; Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Simple Endoscopic Score - Crohn's Disease (SES-CD) | Week 24
  Measuring intestinal health improvement is the Week 24 change from baseline in Simple Endoscopic Score - Crohn's Disease (SES-CD)

SECONDARY OUTCOMES:
Plasma amino acid level | Week 12 and at Week 24
  Change from baseline in plasma amino acid levels
Quality of Life Score - Inflammatory Bowel Disease Questionnaire (IBDQ) | Weeks 12 and 24
  Change from baseline in quality of life score in IBDQ
Quality of Life Score - Work Productivity Activity Index - Crohn's Disease(WPAI-CD) | Weeks 12 and 24
  Change from baseline in quality of life score in WPAI-CD
Inflammatory biomarkers | Week 24
  Proportion of subjects with a normalization of inflammatory biomarkers (C-Reactive Protein (CRP) and fecal calprotectin)
Endoscopic response | Week 24
  Proportion of subjects with endoscopic response based on SES-CD score, defined as a decrease in the SES-CD of at least 3 points from baseline, and no worsening of either component of the PRO2 (abdominal pain or liquid or soft stool frequency)
Corticosteroid-free | Week 12
  Proportion of subjects who are corticosteroid-free

CONTACTS AND LOCATIONS:
Overall Officials: James Lewis, M.D., Study Chair — University of Pennsylvania
Locations (39):
- United States (39):
  - CROWN Site 0032, Dothan, Alabama
  - CROWN Site 0011, Huntsville, Alabama
  - CROWN Site 0091, Little Rock, Arkansas
  - CROWN Site 0017, Los Angeles, California
  - CROWN Site 0054, Rialto, California
  - CROWN Site 0013, Ventura, California
  - CROWN Site 0030, Aurora, Colorado
  - CROWN Site 0028, Bridgeport, Connecticut
  - CROWN Site 0073, Washington D.C., District of Columbia
  - CROWN Site 0096, Naples, Florida
  - CROWN Site 0081, Chicago, Illinois
  - CROWN Site 0050, Urbana, Illinois
  - CROWN Site 0036, Topeka, Kansas
  - CROWN Site 0019, Crestview Hills, Kentucky
  - CROWN Site 0002, Bastrop, Louisiana
  - CROWN Site 0003, Baton Rouge, Louisiana
  - CROWN Site 0029, Shreveport, Louisiana
  - CROWN Site 0051, Chevy Chase, Maryland
  - CROWN Site 0014, Ann Arbor, Michigan
  - Crown Site 0006, Chesterfield, Michigan
  - CROWN Site 71, Lebanon, New Hampshire
  - CROWN Site 0020, Great Neck, New York
  - CROWN Site 0084, Mineola, New York
  - CROWN Site 0039, Poughkeepsie, New York
  - CROWN Site 0012, Asheville, North Carolina
  - CROWN Site 0018, Chapel Hill, North Carolina
  - CROWN Site 0034, Raleigh, North Carolina
  - CROWN Site 0021, Rocky Mount, North Carolina
  - CROWN Site 0093, Portland, Oregon
  - CROWN Site 0033, Philadelphia, Pennsylvania
  - CROWN Site 0040, Philadelphia, Pennsylvania
  - CROWN Site 0094, Rapid City, South Dakota
  - CROWN Site 0041, Hermitage, Tennessee
  - CROWN Site 0004, Houston, Texas
  - CROWN Site 0086, Houston, Texas
  - CROWN Site 0007, Orem, Utah
  - CROWN Site 0016, Norfolk, Virginia
  - CROWN Site 0098, Bellevue, Washington
  - CROWN Site 0009, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No